CLINICAL TRIAL: NCT01629381
Title: Efficacy of RIvaroxaban for Prevention of Venous Thromboembolism After Knee Arthroscopy: a Randomized Double-blind Trial (ERIKA Study)
Brief Title: Efficacy of RIvaroxaban for Prevention of Venous Thromboembolism After Knee Arthroscopy
Acronym: ERIKA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Giuseppe Camporese, MD, Principal Investigator, Coordinator of Emergency Section at the Unit of Angiology, University Hospital of Padua, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2010-024338-43
Record Dates: First submitted 2011-05-09; First posted 2012-06-27 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Venous Thromboembolism; Haemorrhage
Keywords: knee arthroscopy; venous thromboembolism; prevention
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Oral Rivaroxaban 10 mg od for 7 days
  Interventions: Drug: Rivaroxaban
- Placebo (Placebo Comparator): oral placebo od for 7 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rivaroxaban — 10 mg os once daily for 1 week
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: placebo — 10 mg os once daily for 1 week
  Arms: Placebo

SUMMARY:
Study Objective: To assess the value of Rivaroxaban for the prevention of venous thromboembolism (VTE) after knee arthroscopy (KA) taking the placebo as standard of reference.

Study Population: Patients undergoing therapeutic KA at the study Centers, irrespective of the type and duration of the procedure, will be eligible for the study.

Study Design: Multicenter, randomized, double blind superiority, phase II trial comparing two arms:

* (R-7d) Rivaroxaban (10 mg od os) for 7 days
* (PL-7d) Placebo for 7 days.

Follow-up: 3-month period after the randomization

Standard of Reference:Placebo will be the standard of reference in accordance to international guidelines

Study length May 2012-December 2012

Total patients number: 500 patients

Primary Efficacy End-Point: Occurrence in the 3-month period after the randomization of at least one of the following events, objectively proven (by means of CCDU; multi-slice chest TC-angio; autopsy, if necessary, or clinical ground):

* All-cause mortality
* Symptomatic VTE
* Asymptomatic proximal DVT

Secondary Efficacy End-point:

• Combined incidence of all DVT plus symptomatic PE

Primary Safety End-point: Incidence of major bleedings.

Secondary Safety End-point: Overall incidence of bleeding

DETAILED DESCRIPTION:
The treatments will be administered postoperatively (1st dose 8-10 hours after procedure), for prevention of venous thromboembolism after KA.

A bilateral whole-leg colour-coded Doppler ultrasonography (CCDU) is scheduled for all patients at 7 (+1) days of follow-up; additionally, CCDU was due if the patients developed symptoms or signs suggestive of venous thromboembolism earlier.

Statistical & Analytical Plan and Methodology: In the absence of prophylaxis the incidence of venous thromboembolism (primary efficacy end-point) after KA, as assessed by CCDU, is about 8.0% (combining weighted results of various paper). Prophylaxis with low-molecular weight heparins assures approximately a 60-70% relative risk reduction in this setting. Based on the findings of published trials investigating the efficacy of Rivaroxaban for prevention of venous thromboembolism after elective hip and knee surgery, when using a low-molecular-weight heparin as comparator, investigators can speculate that Rivaroxaban will further reduce this incidence (at least 1.2%).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (18 years and older)
2. Knee arthroscopy not combined with open surgery.
3. Patients eligible for surgical treatment.
4. Patients are willing and able to continue study participation to ensure completion of all procedures and observations required by the study.
5. Written informed consent

Exclusion Criteria:

1. Diagnostic arthroscopy
2. Patients concomitantly treated systemically with strong concurrent CYP3A4 and P-gp-inhibitors, i.e. azole-antimycotics or HIV protease inhibitors.
3. Hypersensitivity to the active substance or to any of the excipients of study drug
4. Pregnant women or breast-feeding.
5. Hepatic disease associated with coagulopathy and clinically relevant bleeding risk
6. Known thrombophilia (hereditary or acquired)
7. Mandatory anticoagulation.
8. Known severe bleeding tendency
9. Clinically significant active bleeding.
10. Severe renal failure (GFR<30mL/min/1.73m2)
11. Patients participating in another clinical trial.
12. Recent mayor surgery (6 to 12 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Camporese, MD, Study Chair — Unit of Angiology, University Hospital of Padua, Italy
Locations (9):
- Italy (9):
  - Thrombosis Center & Knee Arthroscopy and Sports Medicine Center, Humanitas Clinical Insitute, Rozzano, Milano
  - Department of Orthopaedics and Traumatology, University Hospital "Galliera" of Genova, Genova
  - Department of Internal Medicine, University Hospital of Napoli, Napoli
  - Department of Orthopaedics and Traumatology, University Hospital of Pavia, Pavia
  - Section of Internal and Cardiovascular Medicine, Department of Internal Medicine, University of Perugia, Perugia
  - Department of Internal Medicine, Hospital of Piacenza, Piacenza
  - Unit of Angiology, Department of Internal Medicine, Azienda Ospedaliera - IRCCS, Reggio Emilia
  - Department of Orthopedics and Surgery of the Hand, Catholic University "Sacro Cuore", Rome
  - Unit of Angiology, Hospital of Venice, Venice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camporese G, Bernardi E, Noventa F, Bosco M, Monteleone G, Santoro L, Bortoluzzi C, Freguja S, Nardin M, Marullo M, Zanon G, Mazzola C, Damiani G, Maniscalco P, Imberti D, Lodigiani C, Becattini C, Tonello C, Agnelli G; ERIKA Study Group. Efficacy of Rivaroxaban for thromboprophylaxis after Knee Arthroscopy (ERIKA). A phase II, multicentre, double-blind, placebo-controlled randomised study. Thromb Haemost. 2016 Aug 1;116(2):349-55. doi: 10.1160/TH16-02-0118. Epub 2016 Apr 14. PMID 27075710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between apr2012 and Mar2014, 1278 subjects were evaluated for inclusion. Of them, 241 (19%) subjects accepted to participate. Due to the unexpectedly low recruitment rate, being a spontaneous study, we were forced to stop the trial before reaching the planned sample size because we were not able to afford insurance costs anymore.
Period: Overall Study
Arm/Group | Rivaroxaban | Placebo
Started | 122 | 119
Completed | 120 | 114
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Placebo | Total
Number analyzed (Participants) | 122 | 119 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.8) | 45.9 (13.9) | 45.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 35 | 79
  Male | 78 | 84 | 162
Region of Enrollment [Number; unit: participants]
  Italy | 122 | 119 | 241

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Symptomatic Venous Thromboembolism Plus Asymptomatic Proximal Vein Thrombosis and All-cause Mortality
Description: During the scheduled visit in case of suspected DVT a bilateral whole-leg colour-coded Doppler ultrasonography (CCDU) is scheduled for all patients at 7 (+1) days of follow-up; additionally, CCDU will be performed if the patients develop symptoms or signs suggestive of venous thromboembolism earlier; in case of suspected PE a multi-slice chest TC-angio is arranged; in case of death for all cause autoptic findings are requested or, if necessary, clinical ground is considered. A follow-up visit is planned 3-month period after the randomization.
Time Frame: 3-month period
Population: Drop-out: seven randomized patients withdrew consent on the day of surgery, without taking the study drug.
Measure: Number; unit: participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 120 | 114
participants | 1 | 7
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority or Other; p = 0.03, Fisher Exact; Risk Difference (RD) = -5.3, 95% CI 2-sided [-11.3 to -0.4]

2. Primary Outcome: Major Bleedings
Description: Major bleeding include: clinically overt haemorrhage associated with haemoglobin drop of at least 2 g/L or requiring the transfusion of two or more units of packed red-blood cells; retroperitoneal or intracranial events; bleeding requiring re-intervention; and hemarthrosis with a joint drainage of more than 450 millilitres of blood.
Time Frame: 3 months
Population: No major bleeding events were observed during the study period.
Measure: Number; unit: participants
Groups:
- Placebo; Rivaroxaban 10 mg for 7 Days: No major bleeding events were observed during the study period.
Arm/Group | Placebo | Rivaroxaban 10 mg for 7 Days
Number analyzed (Participants) | 114 | 120
participants | 0 | 0

3. Secondary Outcome: Combined Incidence of All DVT Plus Symptomatic PE
Description: As described for the assessment of the primary efficacy outcomes
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Placebo: oral placebo od for 7 days placebo: 10 mg os once daily for 1 week
- Rivaroxaban 10 mg for 7 Days: Oral Rivaroxaban 10 mg od for 7 days Rivaroxaban: 10 mg os once daily for 1 week
Arm/Group | Placebo | Rivaroxaban 10 mg for 7 Days
Number analyzed (Participants) | 114 | 120
participants | 8 | 2
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 10 mg for 7 Days; Test type: Superiority or Other; p = 0.03, Fisher Exact; Risk Difference (RD) = -5.3, 95% CI 2-sided [-11.7 to -0.1]

4. Secondary Outcome: Overall Incidence of Bleeding
Description: As described for the primary safety outcome
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Placebo | Rivaroxaban 10 mg for 7 Days
Number analyzed (Participants) | 114 | 120
participants | 6 | 4
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 10 mg for 7 Days; Test type: Superiority or Other; p = 0.53, Fisher Exact; Risk Difference (RD) = -2.0, 95% CI 2-sided [-8.0 to 3.7]

ADVERSE EVENTS:
Time Frame: 7 days on therapy and 90 days of follow-up
Arm/Group | Placebo | Rivaroxaban 10 mg for 7 Days
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/120
Other Adverse Events (participants affected / at risk) | 0/114 | 1/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=114) | Rivaroxaban 10 mg for 7 Days (N=120)
skin reaction (General disorders) | 0 (0) | 1 (1) — spontaneous, moderate, self-recovered skin reaction

LIMITATIONS AND CAVEATS:
Use of placebo instead of active comparator. Small sample size and quite high exclusion rate. Local events adjudication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No